CLINICAL TRIAL: NCT06970730
Title: Evaluation of Accuracy of Virtual Surgical Planning and Patient Specific Implants in Craniomaxillofacial Reconstruction (Clinical Trial)
Brief Title: Accuracy of Virtual Surgical Planning and Patient Specific Implants in Craniomaxillofacial Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Lecturer of Dental Public Health and biostatistical consultanat, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 644-08/2021
Record Dates: First submitted 2025-04-27; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Craniofacial Surgery; Virtual Surgical Planning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- virtual surgical planning and patient specific implants in craniomaxillofacial reconstruction. (Experimental)
  Interventions: Procedure: virtual surgical planning and patient specific implants in craniomaxillofacial reconstruction

INTERVENTIONS:
Procedure: virtual surgical planning and patient specific implants in craniomaxillofacial reconstruction — Image acquisition by computed tomography (CT slice thickness 1 mm or less) + laser scanning of patient models. Virtual surgical planning and design of patient specific implants. Patient specific implants manufacturing (milling technique) and 3D printing of surgical guides and fit models.

SUMMARY:
The sample will consist of 10 patients who will need reconstruction of craniomaxillofacial deformities and defects. The patients will be operated in the Maxillofacial and Plastic Surgery Department, Faculty of Dentistry, Alexandria University, Egypt. All patients will be assessed clinically and radiographically using computed tomography (CT) then virtual surgical planning and custom made patient specific implant will be manufactured. Post-operative clinical evaluation will be done and radiographic evaluation of all patients will be done by CT scan

DETAILED DESCRIPTION:
The primary outcome of the study is to evaluate the accuracy of virtual surgical planning and patient specific implants in craniomaxillofacial reconstruction based on radiographic measurements to calculate the angulation deviations of anatomic landmarks between the pre-operative virtual plan and the post-operative actual surgical outcome.

The secondary outcome is long term follow up of the patients clinically and radiographically regarding aesthetics, quality of life and post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

* Reconstruction of craniofacial, midface, and mandibular bony defects and deformities secondary to:
* Trauma.
* Tumor resection (either by immediate or delayed reconstruction).
* Complex congenital and dentofacial deformities.

Exclusion Criteria:

* Patients with special needs.
* Medically compromised patients who are not fit for surgery.
* Irradiated patients.

Ages: 10 Years to 47 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Distance deviation | Immediate post operative
  the accuracy of reconstruction, defined as linear deviations of anatomic landmarks between the virtual plan and the actual surgical outcome using CT scans
Angular deviation | Immediate post operative
  the accuracy of reconstruction, defined as angulation deviations of anatomic landmarks between the virtual plan and the actual surgical outcome using CT scans

SECONDARY OUTCOMES:
Change in post operative aesthetic results of surgery | 1 week, 4 weeks, 8 weeks, and 6 months
  aesthetic scale from zero to 5
  * 5 points - changes are not visually noticeable.
  * 4 points - changes in appearance are barely noticeable and do not affect the patient's quality of life.
  * 3 points - aesthetic deficit that does not require surgical correction.
  * 2 points - aesthetic defects require minor surgical corrections in the postoperative period.
  * 1 point - significant aesthetic defects require serious (often multi-stage surgical correction).
  * 0 points - the presence of severe aesthetic defects that cannot be eliminated.
change in Quality of Life (QOL) | 1 week, 4 weeks, 8 weeks, and 6 months
  Scores as follow 0 = much better.
  1. = better.
  2. = the same.
  3. = worse.
  4. = much worse

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Azarita, Egypt